CLINICAL TRIAL: NCT02021734
Title: Genetics of Mendelian Diseases in Qatar
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Other Study IDs: 13-00065 [JIRB]; 12217/12 (Other: HMC IRB)
Record Dates: First submitted 2013-11-22; First posted 2013-12-27 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mendelian Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
There are certain categories of diseases which are more prevalent in the Arab world due to increased rates of consanguinity in relatively isolated populations. The goal is to discover these mutations by using next-generation human genetics tools.

DETAILED DESCRIPTION:
There are certain categories of diseases which are more prevalent in the Arab world due to increased rates of consanguinity in relatively isolated populations. The goal is to discover these mutations by using next-generation human genetics tools. These include high-throughput sequencing and genotyping along with the necessary bioinformatics analyses that will lead to the discovery of the causes of most inherited diseases in the region.The secondary objective will be to build a comprehensive catalogue of genetic variation in the Arab world. This will include all detected mutations, not only the subset that are causing disease (from primary objective), but also known trait-altering mutations as well as general diversity on the DNA level among human populations of this region. This catalogue can become a widely useful resource for many projects down the road, as it relies on anonymizing individual samples and instead displaying data in aggregate as the cohorts of collected samples grow over the years.

The study will include all genetic disorders from all ethnic backgrounds but Mendelian disease for which a gene mutation has already been identified will be excluded.

Evidence of Mendelian Transmission determined by fulfilling one of the following criteria:

Multiple affected family members (at least first degree relative with disease) History of consanguinity Severe disease in newborn in the absence of family history Sydromic disease in single individuals Congenital abnormality affecting major organ system(s) Mendelianized extremes of common disease (eg sever familial diabetes/ obesity/ hypertension)

ELIGIBILITY:
Inclusion Criteria:

* All included individuals must provide informed consent
* All genetic disorders are included
* All ethnic backgrounds are accepted
* Disease must be genetic with no evident environmental cause
* Evidence of Mendelian Transmission determined by fulfilling one of the following criteria:
* Multiple affected family members (at least first degree relative with disease)
* History of consanguinity
* Severe disease in newborn in the absence of family history
* Sydromic disease in single individuals
* Congenital abnormality affecting major organ system(s)
* Mendelianized extremes of common disease (eg sever familial diabetes/ obesity/ hypertension)

Exclusion Criteria:

* Individuals who do no consent to be included
* Mendelian disease for which a gene mutation has already been identified
* Individuals for which a molecular diagnosis has already been established by alternative method
* Disease for which an environmental factor is most likely the cause
* Disease for which late age of onset rule out Mendelian transmission
* Common diseases for which late age of onset rule out Mendelian transmission

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: physicians and by thorough review of the literature to establish that the disease is indeed Mendelian and with unknown gene.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-11-19 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2025-02 (Actual)

PRIMARY OUTCOMES:
Next generation sequencing | 1 hour
  Use next generation sequencing to detect novel disease causing mutations

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No